CLINICAL TRIAL: NCT04004364
Title: Early-Phase Schizophrenia: Practice-based Research to Improve Outcomes
Acronym: ESPRITO
Status: Recruiting | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: ESPRITO 19-0307
Record Dates: First submitted 2019-06-28; First posted 2019-07-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: First Episode Psychosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Coordinated Specialty Care (CSC) — CSC is an integrated and team-based treatment model for first episode psychosis elements include psychotherapy, supported employment and education, family education and support, and pharmacotherapy.

SUMMARY:
The goal if the project is to develop a learning health network devoted to the treatment of first episode psychosis.

DETAILED DESCRIPTION:
The RAISE ETP study, designed and conducted by our group, signaled that a Coordinated Specialty Care (CSC) model could be feasibly delivered in community mental health clinics in multiple states and was effective. Since then, with the support of SAMSHA block grants to states, there are CSC programs across the nation.

The goal of this project is to develop a learning health system with sites providing CSC treatment of first-episode psychosis (FEP). Sites are drawn from five states: Connecticut, Florida, Michigan, Oklahoma and South Carolina. They vary in populations served, levels of funding available and research experience. All are committed to advancing the development of CSC using a health learning system model, to implementing a practical assessment strategy to enhance outcome assessment and to conducting research to improve outcomes that will be meaningful to the full range of stakeholders.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in CSC program

Exclusion Criteria:

* none

Ages: 15 Years to 40 Years | Sex: All
Age Groups: Child, Adult
Study Population: 15 to 40 year olds with first episode psychosis enrolled in network CSC program
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of Enrolled participants | 5 years of the project
  Number of enrolled participants into the learning health system

CONTACTS AND LOCATIONS:
Locations (1):
- Henderson Behavioral Health, Lauderdale Lakes, Florida, United States

IPD SHARING:
Plan to Share IPD: No